CLINICAL TRIAL: NCT02088112
Title: A Phase I, Open-Label, Multicentre Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumour Activity of Gefitinib in Combination With MEDI4736 (Anti PD-L1) in Subjects With Non-Small Cell Lung Cancer(NSCLC)
Brief Title: MEDI4736 (Anti PD-L1) Combined With Gefitinib in Subjects With Non-Small Cell Lung Cancer(NSCLC).
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D791PC00001
Record Dates: First submitted 2014-03-07; First posted 2014-03-14 (Estimated); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Escalation (Experimental): MEDI4736 will be combined with gefitinib to assess safety and tolerability
  Interventions: Drug: Gefitinib; Drug: MEDI4736
- Expansion Arm (Experimental): MEDI4736 will be combined with gefitinib
  Interventions: Drug: Gefitinib; Drug: MEDI4736

INTERVENTIONS:
Drug: Gefitinib — Gefitinib QD
Drug: MEDI4736 — MEDI4736 IV Q2W

SUMMARY:
This a Phase I, Open-Label, Multicentre Study to assess the safety, tolerability, pharmacokinetics and preliminary anti-tumour activity of gefitinib in combination with MEDI4736 (anti PD-L1) in Subjects with Non-small cell lung cancer (NSCLC). The study consists of two phases: Escalation phase and an expansion phase to be conducted in locally advanced or metastatic NSCLC subjects

DETAILED DESCRIPTION:
In Escalation phase: MEDI4736 and gefitinib in NSCLC subjects In Expansion phase: Subjects with EGFR mutation positive locally advanced or metastatic NSCLC will be enrolled in expansion arms. Initiation of expansion arms with the recommended dose of MEDI4736 in combination with gefitinib will be based on an adequate safety and tolerability profile of the combination from the escalation phase.

ELIGIBILITY:
Key Inclusion Criteria:

1. Provision of signed and dated, written informed consent
2. Male or female aged 18 years and older.
3. Subjects must have a. In the escalation phase, locally advanced or metastatic NSCLC subjects who have either failed to respond or relapsed following any line of standard treatment, were unable to tolerate, or were not eligible for standard treatment b. In the expansion phase, histologically or cytologically confirmed locally advanced or metastatic NSCLC that is EGFR mutation positive, naïve to EGFR TKI therapy, and sensitive to EGFR TKIs therapy
4. a.For Escalation Phase: At least one lesion (measurable and/or non-measurable) b.For Expansion Phase: At least one measurable lesion.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

   * For Japan Escalation - the same as the global escalation I/E criteria except patients must be EGFR mutation positive

Key Exclusion Criteria:

1. Any concurrent chemotherapy, immunotherapy, biologic, or hormonal therapy for cancer treatment.
2. Any investigational agent, chemotherapy, immunotherapy, biologic, hormonal within 28 days of the first dose of study treatment
3. Inadequate bone marrow reserve or organ function

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2014-03-24 (Actual); Primary Completion 2021-03-09 (Actual); Study Completion 2021-03-09 (Actual)

PRIMARY OUTCOMES:
Escalation Phase: safety and tolerability: AEs, laboratory data, vital signs, ECG changes and Echo. Expansion Phase: safety and tolerability of the recommended dose for MEDI4736; AEs, laboratory data, vital signs, ECG changes and Echo. | From first dose of study treatment until 90 days after the last dose, assessed up to 32 months
  AEs: Type, incidence, severity, seriousness and relationship to study medications of adverse events (AE) (graded by the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE]; Safety Labs: Blood and urine samples for determination of clinical chemistry, hematology, coagulation, thyroid function tests and urinalysis will be taken at the visits; any laboratory abnormalities, and including dose-limiting toxicities (DLTs), ECG measurements and Creatinine Clearance

SECONDARY OUTCOMES:
To obtain a preliminary assessment of the anti-tumour activity of gefitinib in combination with MEDI4736 by evaluation of tumour response | From baseline assessment to disease progression, assessed up to 30 months
  At each visit subjects will be programmatically assigned a RECIST visit response of CR, PR, SD or PD depending on the status of their disease compared to baseline and previous assessments; Objective response rate: the percentage of subjects who have at least one visit response of CR or PR prior to any evidence of progression . Disease control rate: the percentage of subjects who have at least one visit response of CR or PR or SD prior to any evidence of progression. Progression Free Survival (PFS) : the time from start of study treatment to the first documentation of objective disease progression (PD) or death from any cause.
To determine the immunogenicity of MEDI4736 in combination with gefitinib: anti-drug antibodies (ADAs) | From first dose of study treatment until 90 days after the last dose, assessed up to 32 months
  Assessed by evaluating the number and percentage of subjects who develop detectable anti-drug antibodies (ADAs). The impact of ADAs on overall MEDI4736 PK will also be evaluated.
To determine the pharmacokinetics of MEDI4736 | From first dose of study treatment until 90 days after the last dose, assessed up to 32 months
  Individual MEDI4736 concentrations will be tabulated by dose cohort along with descriptive statistics. Noncompartmental PK data analysis will be performed
To assess MEDI4736 pharmacodynamics in subjects receiving MEDI4736 in combination with gefitinib. | From first dose of study treatment until 90 days after the last dose, assessed up to 32 months
  PD-L1 levels before and after treatment with MEDI4736 will be measured to evaluate its association with response to treatment with MEDI4736 and clinical outcome
To determine overall survival (OS) in expansion Arm 1 and Arm 1a patients | From final safety follow-up visit after last dose until 1 year after the final patient discontinues investigational product (initial Medi4736).
  Survival information may be obtained via telephone contact with the patient, patients family or by checking the patients notes, hospital records, contacting the patients general practitioner or public death registry, where it is possible to do so under applicable local laws.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Creelan, MD, Principal Investigator — Moffit Cancer Center; Don Gibbons, MD, Principal Investigator — M.D. Anderson Cancer Center; Laura Chow, MD, Principal Investigator — University of Washington; Sang-We Kim, MD, Principal Investigator — Asan Medical Center; Dong-Wan Kim, MD, Principal Investigator — Seoul National University Hospital; Shinitaro Kanda, MD, Principal Investigator — National Cancer Center; Naoyuki Nogami, Principal Investigator — Shikoku Cancer Center
Locations (6):
- United States (3):
  - Research Site, Tampa, Florida
  - Research Site, Houston, Texas
  - Research Site, Seattle, Washington
- Japan (2):
  - Research Site, Chūōku
  - Research Site, Matsuyama
- Research Site, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Creelan BC, Yeh TC, Kim SW, Nogami N, Kim DW, Chow LQM, Kanda S, Taylor R, Tang W, Tang M, Angell HK, Roudier MP, Marotti M, Gibbons DL. A Phase 1 study of gefitinib combined with durvalumab in EGFR TKI-naive patients with EGFR mutation-positive locally advanced/metastatic non-small-cell lung cancer. Br J Cancer. 2021 Jan;124(2):383-390. doi: 10.1038/s41416-020-01099-7. Epub 2020 Oct 5. PMID 33012782
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D791PC00001&attachmentIdentifier=6d02987f-bf7f-4ce3-b7ef-21a80cb1c46e&fileName=d791pc00001-study-CSR_synopsis_Redacted_14Jan2022.pdf&versionIdentifier=
- See also: Results of this clinical trial are available on www.astrazenecaclinicaltrials.com — https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Search